CLINICAL TRIAL: NCT01393210
Title: The Influence of Beta-glucan 1.3D-1.6D, Added to the Low-calorie Diet, on Insulin Sensitivity and the Expression of Selected Proinflammatory Cytokines in Adipose Tissue and Peripheral Blood Mononuclear Cells in Obese Humans
Brief Title: Beta-glucan and Insulin Sensitivity in Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marek Straczkowski (Other)
Responsible Party: Sponsor-Investigator, Marek Straczkowski, Prof., Polish Academy of Sciences
Organization: Polish Academy of Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPChM-11-01
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: insulin sensitivity; adipose tissue; inflammation
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation | interventions — Caloric Restriction; beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-calorie diet (Active Comparator): Intervention was low-calorie diet only for 12 weeks.
  Interventions: Other: low-calorie diet
- low calorie diet plus beta-glucan (Active Comparator): Intervention was low-calorie diet plus BETA-GlLUCAN 1.3D-1.6D 500 mg daily for 12 weeks.
  Interventions: Dietary Supplement: low calorie diet plus beta-glucan; Other: low-calorie diet

INTERVENTIONS:
Dietary Supplement: low calorie diet plus beta-glucan — beta-glucan 1.3D-1.6D, together with a low calorie diet, 500 mg once daily for 12 weeks
  Arms: low calorie diet plus beta-glucan
Other: low-calorie diet — low-calorie diet only for 12 weeks.

SUMMARY:
Obesity is an important health problem of modern civilization. In Western societies, almost half of the adult population has problems with an increased body weight. Products containing nutritional fiber has been used by humans for thousands of years. However, beta-glucan as biologically active compound, present in these products, has been identified relatively lately. This substance is a polymer of glucose and is present in two forms: 1,3D-1,6D and 1,3D-1,4D.

Water-insoluble beta-glucan (1,3D-1,6D) has immunomodulatory properties. The aim of the study was the assessment of the influence of beta-glucan 1,3D-1,6D added to the low-calorie diet on insulin sensitivity and the expression of selected proinflammatory cytokines in adipose tissue and peripheral blood mononuclear cells (PBMC) in obese humans with normal glucose tolerance.

The study group consisted of 40 subjects with marked overweight or obesity (body mass index, BMI > 28 kg/m2), without serious concomitant diseases not taking drugs affecting glucose or lipid metabolism, nonsmokers. Only volunteers, who gave written informed consent, after receiving a full information about the aim and the design of the study, were recruited.

At the beginning of the study, after subjects' qualification to the project and before the dietary intervention, the investigators performed:

* anthropometric measurements.
* oral glucose tolerance test.
* euglycemic hyperinsulinemic clamp.
* PBMC isolation before and after the clamp.
* biopsy of subcutaneous adipose tissue before the clamp.
* isolation of mRNA from PBMC and adipose tissue. Then, the expression of the selected genes with the Real Time PCR was measured.
* After the initial visit, participants received detailed instructions about low-calorie diet, with the aim of reduction of 5-7% of body weight and the examples of menu for 14 days.

Then, participants were randomly assigned to a group receiving or not beta-glucan preparation, as a addition to the low-calorie diet. Each group consisted of 20 subjects. Subjects assigned to a group receiving beta-glucan, received the preparation (BETA GLUCAN 1,3-1,6 Laboratoria Natury 500mg) together with the detailed instruction of its usage. This preparation is used as a non-prescription diet supplement, and the dose of 500 mg daily is indicated by the manufacturer.

After 12 weeks of low-calorie diet, without or with beta-glucan, all the examinations performed at the beginning of the study were repeated.

DETAILED DESCRIPTION:
Obesity is an important health problem of modern civilization. In Western societies, almost half of the adult population has problems with an increased body weight. In Europe, obesity occurs in 10-20% males and 15-25% females. In Poland, obesity is present in about 20% of population.

Products containing nutritional fiber has been used by humans for thousands of years. However, beta-glucan as biologically active compound, present in these products, has been identified relatively lately. This substance is a polymer of glucose and is present in two forms: 1,3D-1,6D and 1,3D-1,4D.

Water-insoluble beta-glucan (1,3D-1,6D) has immunomodulatory properties. It stimulates host defense against viral, bacterial and parasitical infections through binding with the specific receptors located on the immune system cells surface in many animal models. There are data that beta-glucan 1,3D-1,6D affects both innate and acquired immune response also in humans.

The aim of the study was the assessment of the influence of beta-glucan 1,3D-1,6D added to the low-calorie diet on insulin sensitivity and the expression of selected proinflammatory cytokines in adipose tissue and peripheral blood mononuclear cells (PBMC) in obese humans with normal glucose tolerance.

The study group consisted of 40 subjects with marked overweight or obesity (body mass index, BMI > 28 kg/m2), without serious concomitant diseases not taking drugs affecting glucose or lipid metabolism, nonsmokers. Only volunteers, who gave written informed consent, after receiving a full information about the aim and the design of the study by the research personnel were recruited.

At the beginning of the study, after subjects' qualification to the project and before the dietary intervention, the investigators assessed:

* anthropometric measurements: BMI, waist-to-hip ratio (WHR), full physical examination.
* body composition with Tanita TBF-511 Body Fat Analyzer.
* glucose tolerance with the oral glucose tolerance test.
* insulin sensitivity with the euglycemic hyperinsulinemic clamp technique.
* before and after the clamp, additional 6 ml of blood was collected, and PBMC isolation was performed.
* before the clamp, a biopsy of subcutaneous adipose tissue was performed.
* isolation of mRNA from PBMC and adipose tissue was performed. Then, the expression of the selected genes with the Real Time PCR In adipose tissue was measured measured.
* additionally, serum concentrations of ghrelin, peptide Y-Y3-36, citruline and intestinal fatty acid-binding protein was assessed.

After the initial visit, participants received detailed instructions about low-calorie diet, with the aim of reduction of 5-7% of body weight and the examples of menu for 14 days.

Then, participants were randomly assigned to a group receiving or not beta-glucan preparation, as a addition to the low-calorie diet. Each group consisted of 20 subjects. Subjects assigned to a group receiving beta-glucan, received the preparation (BETA GLUCAN 1,3-1,6 Laboratoria Natury 500mg) together with the detailed instruction of its usage. This preparation is used as a non-prescription diet supplement, and the dose of 500 mg daily is indicated by the manufacturer.

Analysis of the compliance to the dietary indications and analysis of body composition was performed every 2 weeks.

After 12 weeks of low-calorie diet, without or with beta-glucan, all the examinations performed at the beginning of the study were repeated.

ELIGIBILITY:
Inclusion Criteria:

* marked overweight or obesity (BMI above 28 kg/m2)
* normal glucose tolerance

Exclusion Criteria:

* morbid obesity (BMI above 40 kg/m2)
* impaired glucose tolerance or diabetes
* cardiovascular diseases
* other serious disease
* smoking
* usage of drugs known to affect carbohydrate or lipid metabolism

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | one year

SECONDARY OUTCOMES:
body weight | one year
amount of visceral adipose tissue | one year
expression of selected genes in PBMC and adipose tissue | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marek Straczkowski, MD, prof., Principal Investigator — Institute of Animal Reproduction and Food Research, Polish Academy of Sciences
Locations (1):
- Institute of Animal Reproduction and Food Research, Polish Academy of Sciences, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danowska M, Stefanowicz M, Straczkowski M. The expression of NFAT family genes in subcutaneous adipose tissue before and after weight loss in obese individuals. Nutr Metab Cardiovasc Dis. 2024 Nov;34(11):2455-2463. doi: 10.1016/j.numecd.2024.06.011. Epub 2024 Jun 20. PMID 39069466
- [Derived] Nikolajuk A, Stefanowicz M, Straczkowski M, Karczewska-Kupczewska M. Changes in Adipose Tissue Gene Expression of the Core Components of the Hippo Signaling Pathway in Young Adults with Uncomplicated Overweight or Obesity Following Weight Loss. J Nutr. 2023 Mar;153(3):665-672. doi: 10.1016/j.tjnut.2023.01.024. Epub 2023 Jan 26. PMID 36805181